CLINICAL TRIAL: NCT06456775
Title: Tele-SSM: A Telephone Technology Innovation in the Intervention on Supported Self-management for Depression in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Social Development Studies, Vietnam (Other)
Collaborators: National Foundation for Science & Technology Development, Vietnam (Unknown)
Responsible Party: Principal Investigator, Tran Kieu Nhu, Head of Research Division, Institute for Social Development Studies, Vietnam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NCUD.05-2019.29
Record Dates: First submitted 2024-06-05; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Depression
Keywords: depression; supported self-management; task-shifting approach; mobile health; mental health; Vietnam
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Single Group: Clinical trials with a single arm
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): All participants in the study received a supported self-management intervention for depression delivered from distance.
  Interventions: Behavioral: Tele-SSM

INTERVENTIONS:
Behavioral: Tele-SSM — Tele-SSM an individual-level psychosocial intervention based on cognitive behavior therapy principles and non-violent communication. The intervention consists of the following 10 sessions delivered through 10 weekly coaching calls delivered by Zoom (audio only).

SUMMARY:
Tele-SSM is a pre-post mixed-method study to investigate the feasibility, acceptability and the preliminary efficacy of the support self-management skills intervention for depression delivered from distance.

The specific objectives of this research include:

* Transform the SSM intervention for depression from face-to-face delivery to delivery from distance.
* Develop an software for intervention management
* Examine knowledge, attitudes and practices of people with depression toward depression
* Examine the feasibility, acceptability and preliminary efficacy of the intervention
* Investigate the cost analysis of Tele-SSM intervention

DETAILED DESCRIPTION:
Introduction

In the context of limited interventions for depression in Vietnam and the strong potential for tele-health to improve accessibility to mental health care in low-middle income countries, the principal investigators conducted a pre-post mixed-method study of a supported self-management for depression delivered from distance (Tele-SSM) to evaluate the preliminary efficacy, feasibility and acceptability of this approach on depression and other mental health outcomes for adults with depression symptoms in Vietnam and to explore knowledge, attitudes and practices of people with depression towards depression.

Method

This is pre-post mixed method study. The princial investigators use both quantitative and quanlitative methodology to evaluate the preliminary efficacy, feasibility and acceptability of Tele-SSM intervention on depression and other mental health outcomes for adults with depression symptoms in Vietnam and to explore knowledge, attitudes and practices of people with depression towards depression.

Recruitment

Participants ages 18-64 years ared recruited online through social media from May 2022 and May 2023. Interested participants completed the PHQ-9 on Kobotoolbox. Potential participants who satisfy the eligibility criteria of the study provided contact information. A research assistant with a psychology background conducted a video call with each potential participant to confirm their eligibility, provide information about the study and the intervention. Informed consent was obtained from all individual participants included in the study.

All procedures performed in studies involving human participants are in accordance with the ethical standards of the institutional ethical committee and was approved by the Institutional Review Board at ISDS (IRB00011703) on 05th May 2021 in Hanoi.

Sample size considerations

Findings from meta-analytic studies examining the effect of CBT interventions indicate the effect size for CBT on depressive symptoms to be 0.53 (Cuijpers et al., 2013) and on health-related quality of life to be 0.63 (Hofmann et al., 2017). Sample size calculations indicated that a sample size of 52 participants was sufficient to detect a conservative anticipated effect size of 0.40, with a statistical power of 80% and a two-sided alpha level of 0.05. The target sample size was increased to 72, assuming an anticipated attrition rate of 20%. In reality, the principal investigators recruited 75 patients, with 58 patients completing the intervention.

Data management

* Participants completed pre- and post-questionnaires online using Kobotoolbox. The in-depth interviews are audio-recorded. Audio recordings are transcribed. Participant records are managed by a secured website.

Data Analysis Plan

* Qualitative analysis methods: The IDIs are audio-recorded, transcribed and analyzed thematically to identify significant themes, patterns, and potential correlational relationships. The analysis is conducted with Excel software.
* Quantitative analysis method: The principal investigators calculate descriptive statistics for all variables (means, ranges, standard deviations, percent data missing, and frequencies for categorical variables). For continuous variables, the principal investigators conduct statiscial tests to test for differences before and after intervention. For the acceptability, frequencies for questions on satisfaction were calculated from endline data.
* Cost analysis method: The principal investigators analyze all costs incurred from activities of Tele-SSM intervention for all participants in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged from 18-64 years
* Have a score of PHQ-9 (26) greater than 5.

Exclusion Criteria:

* Any participants with severe mental health problems i.e. schizophrenia, bipolar disorder, recent suicide attempts and/or with suicide plans were excluded (current suicide ideation, but without recent suicide attempts and/or with suicide plans were not excluded).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Depression | Pre intervention and up to 12 weeks
  Measured by PHQ-9 questionnaire
Acceptability | Up to 12 weeks after pre-intervention survey
  Measured by questionnaire and in-depth interviews
Feasiblity | Up to 12 weeks after pre-intervention survey
  Measured by questionnaire and in-depth interviews
Cost | Through study completion, an average 6 months
  Measured by financial reports

SECONDARY OUTCOMES:
Anxiety | Pre intervention and up to 12 weeks
  Measure by DASS-21 questionnaire
Stress | Pre intervention and up to 12 weeks
  Measured by DASS-21 questionnaire
Self-esteem | Pre intervention and up to 12 weeks
  Measured by Rosenberg self - Esteem scale
Social support | Pre intervention and up to 12 weeks
  Measured by Multidimensional Scale of Perceived Social Support (MSPSS)
Health related quality of life | Pre intervention and up to 12 weeks
  Measured by SF-12 and EQ-5D-5L questionnaire
Knowledge, attitude and practices of people with depression | Pre-intervention
  Measured by in-depth interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Social Development Studies, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The data of this study are available on request from the principal investigator after the outcomes of the study are published. .
Supporting Information: SAP, ICF, CSR
Time Frame: The data is available upon request after the outcomes of the study are published.
Access Criteria: Researchers must sign a Data Use Agreement specifying the terms and conditions of data usage, including confidentiality, data security measures, and prohibitions on unauthorized data sharing. Researchers must be affiliated with a recognized academic, governmental, or non-profit research institution.
  Proof of institutional affiliation may be required.esearchers must adhere to ethical guidelines and legal regulations governing data protection and privacy. Data should be used for the purposes outlined in the approved agreement.

REFERENCES:
- [Background] Konig H, Konig HH, Konnopka A. The excess costs of depression: a systematic review and meta-analysis. Epidemiol Psychiatr Sci. 2019 Apr 5;29:e30. doi: 10.1017/S2045796019000180. PMID 30947759
- [Background] Christensen MK, Lim CCW, Saha S, Plana-Ripoll O, Cannon D, Presley F, Weye N, Momen NC, Whiteford HA, Iburg KM, McGrath JJ. The cost of mental disorders: a systematic review. Epidemiol Psychiatr Sci. 2020 Aug 18;29:e161. doi: 10.1017/S204579602000075X. PMID 32807256
- [Background] Cuijpers P, Noma H, Karyotaki E, Cipriani A, Furukawa TA. Effectiveness and Acceptability of Cognitive Behavior Therapy Delivery Formats in Adults With Depression: A Network Meta-analysis. JAMA Psychiatry. 2019 Jul 1;76(7):700-707. doi: 10.1001/jamapsychiatry.2019.0268. PMID 30994877
- [Background] Cuijpers P, Karyotaki E, Reijnders M, Purgato M, Barbui C. Psychotherapies for depression in low- and middle-income countries: a meta-analysis. World Psychiatry. 2018 Feb;17(1):90-101. doi: 10.1002/wps.20493. PMID 29352530
- [Background] Bilsker D, Goldner EM, Anderson E. Supported self-management: a simple, effective way to improve depression care. Can J Psychiatry. 2012 Apr;57(4):203-9. doi: 10.1177/070674371205700402. PMID 22480584
- [Background] Linde K, Sigterman K, Kriston L, Rucker G, Jamil S, Meissner K, Schneider A. Effectiveness of psychological treatments for depressive disorders in primary care: systematic review and meta-analysis. Ann Fam Med. 2015 Jan-Feb;13(1):56-68. doi: 10.1370/afm.1719. PMID 25583894
- [Background] Pasarelu CR, Andersson G, Bergman Nordgren L, Dobrean A. Internet-delivered transdiagnostic and tailored cognitive behavioral therapy for anxiety and depression: a systematic review and meta-analysis of randomized controlled trials. Cogn Behav Ther. 2017 Jan;46(1):1-28. doi: 10.1080/16506073.2016.1231219. Epub 2016 Oct 7. PMID 27712544
- [Background] Chau LW, Murphy J, Nguyen VC, Lou H, Khanh H, Thu T, Minas H, O'Neil J. Lay social workers implementing a task-sharing approach to managing depression in Vietnam. Int J Ment Health Syst. 2021 May 29;15(1):52. doi: 10.1186/s13033-021-00478-8. PMID 34051848
- [Background] Connolly SM, Vanchu-Orosco M, Warner J, Seidi PA, Edwards J, Boath E, Irgens AC. Mental health interventions by lay counsellors: a systematic review and meta-analysis. Bull World Health Organ. 2021 Aug 1;99(8):572-582. doi: 10.2471/BLT.20.269050. Epub 2021 Apr 29. PMID 34354312
- [Background] Murphy JK, Xie H, Nguyen VC, Chau LW, Oanh PT, Nhu TK, O'Neil J, Goldsmith CH, Van Hoi N, Ma Y, Lou H, Jones W, Minas H. Is supported self-management for depression effective for adults in community-based settings in Vietnam?: a modified stepped-wedge cluster randomized controlled trial. Int J Ment Health Syst. 2020 Feb 12;14:8. doi: 10.1186/s13033-020-00342-1. eCollection 2020. PMID 32071614
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Background] Murphy J, Goldsmith CH, Jones W, Oanh PT, Nguyen VC. The effectiveness of a Supported Self-management task-shifting intervention for adult depression in Vietnam communities: study protocol for a randomized controlled trial. Trials. 2017 May 5;18(1):209. doi: 10.1186/s13063-017-1924-5. PMID 28476148
- [Derived] Tran NK, Ngo TT, Nguyen TK, Murphy JK, Dang HM. Feasibility, acceptability, and preliminary efficacy of a telehealth supported self-management intervention for adults with depression symptoms in Vietnam: a mixed-method pre-post study. Pilot Feasibility Stud. 2025 Dec 10;12(1):8. doi: 10.1186/s40814-025-01750-1. PMID 41372992
- [Derived] Tran NK, Nguyen QT, Nguyen TK, Hoang MV, Kane S, Dang HM. Knowledge, attitudes, and practices toward depression among people living with depression in Vietnam: the cultural dynamics in the era of globalization. BMC Psychol. 2025 Aug 29;13(1):983. doi: 10.1186/s40359-025-03281-z. PMID 40883799
- Available data/document: Individual Participant Data Set — https://bit.ly/49RBPuQ